CLINICAL TRIAL: NCT06409169
Title: Dried Blood Spot Testing in Peer-assisted Telemedicine for Hepatitis C Treatment
Brief Title: DBS TaT in Peer-assisted Telemedicine for Hepatitis C
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); Oregon Clinical and Translational Research Institute (Other); Collins Medical Trust (Other)
Responsible Party: Principal Investigator, Hunter Spencer, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00026983; KL2TR002370 (NIH)
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Substance Use
MeSH Terms: conditions — Hepatitis C; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DBS TaT (Experimental): At DBS TaT sites, peers administer dried blood spot tests to all those interested in HCV screening or treatment. When HCV is diagnosed, peers coordinate a telemedicine visit with a PATHS provider and peer. At the time of the telemedicine visit, a questionnaire, Decompensated Cirrhosis in Hepatitis C Evaluation Questionnaire (DCHEQ), is used to determine risk level of liver fibrosis (liver scaring that is sometimes caused by hepatitis C). Those at low risk for liver fibrosis can start HCV treatment before completing the usual tests for liver fibrosis. Those at high risk for liver fibrosis will be directed to receive a confirmatory blood draw at a local laboratory prior to treatment initiation. Participants will complete transient elastography after treatment initiation.
  Interventions: Other: DBS TaT
- Usual Care (Active Comparator): At usual care sites, participants either self-report a known history of untreated HCV or undergo peer-performed point-of-care HCV antibody testing or DBS for HCV testing. Peers take those with positive results to local laboratories for a confirmatory blood draw prior to treatment initiation, the results of which are received and managed by PATHS providers. When active HCV is diagnosed, PATHS staff coordinate on-demand telemedicine visits with peers and participants, during which PATHS clinicians recommend treatment. Participants will complete transient elastography after treatment initiation.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: DBS TaT — Dried Blood Spot (DBS) testing for HCV DCHEQ and Baseline Surveys If at high risk for liver fibrosis, blood draw prior to treatment initiation If low risk for liver fibrosis, Telemedicine visit with PATHS provider HCV treatment initiation Transient elastography (TEG)
  Arms: DBS TaT
Other: Usual Care — Point-of-care or DBS testing for HCV Blood draw to test liver fibrosis DCHEQ and Baseline Surveys Telemedicine visit with PATHS provider HCV treatment initiation Transient elastography (TEG)
  Arms: Usual Care

SUMMARY:
The purpose of this study is to compare the rate of treatment initiation achieved by peer-assisted telemedicine contingent on phlebotomy (usual care) versus that achieved with a new protocol, called Dried Blood Spot Test and Treat (DBS TaT). DBS TaT includes DBS testing to diagnose hepatitis C (HCV), utilizes a novel clinical decision aid that identifies patients who are low risk for hepatic (liver) fibrosis, and directs those patients to HCV treatment initiation prior to routine hepatic fibrosis assessment.

The investigators hypothesize that DBS TaT will increase the rate of HCV treatment initiation compared to peer-assisted telemedicine contingent on phlebotomy (usual care).

DETAILED DESCRIPTION:
Oregon has the fourth highest prevalence of hepatitis C (HCV) and third highest HCV-related mortality in the nation and it predominantly effects people who use drugs (PWUD). To respond to this, Peer Assisted Telemedicine for Hepatitis C (PATHS), a Substance Abuse and Mental Health Services Administration supported telemedicine-based HCV treatment program that serve PWUD in predominantly rural areas of Oregon was created. PATHS partners with "peers," people with lived experience of substance use, who work for community-based organizations serving PWUD in high-needs rural counties. Patients are referred to PATHS from opiate treatment programs and community-based organizations throughout the state, which are PATHS' "sites."

The leading barrier to HCV treatment initiation within PATHS is the requirement for participants to complete phlebotomy prior to treatment. To address this problem, PATHS is piloting the use of commercially available, laboratory-validated dried blood spot (DBS) tests to confirm active HCV, but patients who complete DBS must still undergo either phlebotomy or transient elastography (TEG) to complete guideline-recommended hepatic fibrosis staging before HCV treatment. Transient elastography is a validated, non-invasive, clinical standard of hepatic fibrosis assessment covered by Oregon Medicaid, but it is inconvenient to access in rural areas.

This study aims to determine the impact of Dried Blood Spot Test and Treat (DBS TaT) compared to phlebotomy-contingent treatment (usual care) in a cluster randomized controlled trial performed within Peer Assisted Telemedicine for Hepatitis C (PATHS). The primary outcome is the rate of treatment initiation in PATHS sites utilizing DBS TaT versus PATHS sites utilizing usual care. 18 PATHS sites are randomized to DBS TaT implementation or ongoing usual care. Within DBS TaT, participants with low risk for hepatic fibrosis will be offered HCV treatment without phlebotomy but will still undergo imaging-based hepatic fibrosis assessment to ensure safety.

ELIGIBILITY:
Inclusion Criteria:

* Active hepatitis C infection
* Willing to engaged with the PATHS program for clinical care

Exclusion Criteria:

• Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
HCV Treatment Initiation | 12 weeks after diagnosis of HCV
  Rate of hepatitis C (HCV) treatment initiation in sites utilizing DBS TaT versus sites utilizing usual care.

SECONDARY OUTCOMES:
HCV Cure | 24 weeks after treatment completion
  Rate of hepatitis C (HCV) cure in sites utilizing DBS TaT versus sites utilizing usual care tested within 24 weeks of treatment initiation.
Time from HCV Diagnosis to Treatment Initiation | 12 weeks
  Time from diagnosis of HCV to HCV treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Hunter Spencer, DO, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No